CLINICAL TRIAL: NCT04654403
Title: Phase II Study of First-line Camrelizumab With or Without Chemotherapy for Advanced Esophageal Squamous Cell Cancer
Brief Title: Study of First-line Camrelizumab With or Without Chemotherapy for Advanced Esophageal Squamous Cell Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Director, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR1210-016
Record Dates: First submitted 2020-11-19; First posted 2020-12-04 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Esophageal Cancer
Keywords: Advanced or metastatic esophageal squamous cell cancer(ESCC)
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab (Experimental): Camrelizumab (200 mg every 2 weeks),Treatment will continue until confirmed radiographic progression,unacceptable toxicity, investigator or patient decision to withdraw, nonadherence to treatment or trial procedures or completion of 16 cycles of Camrelizumab (approximately 1 years)
  Interventions: Drug: Camrelizumab
- Camrelizumab plus chemotherapy (Active Comparator): Camrelizumab plus chemotherapy(Camrelizumab 200 mg every 3 weeks,docetaxel 75mg/m2/d plus cisplatin 75 mg/m2/d on day 1 every 3 weeks),)Treatment will continue until confirmed radiographic progression,unacceptable toxicity, investigator or patient decision to withdraw, nonadherence to treatment or trial procedures or completion of 16 cycles of Camrelizumab (approximately 1 years).
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Eligible patients receive Camrelizumab 200 mg by intravenous (iv.) infusion every 2 weeks (Q2W) for 4 cycles.Imaging will be performed 2-3 weeks after the 4th Camrelizumab administration.Patients who achieve PD and SD will be not included in the data statistics of this trial.The follow-up treatment according to investigator's and patients's choice(chemotherapy, Camrelizumab plus chemotherapy or Camrelizumab monotherapy).Other patients whose BOR is in remission (CR+PR) will be randomly assigned in a 1:1 ratio to receive Camrelizumab (200 mg every 2 weeks), or Camrelizumab plus chemotherapy(Camrelizumab 200 mg every 3 weeks,docetaxel 75mg/m2/d plus cisplatin 75 mg/m2/d on day 1 every 3 weeks),)Treatment will continue until confirmed radiographic progression,unacceptable toxicity, investigator or patient decision to withdraw, nonadherence to treatment or trial procedures or completion of 16 cycles of Camrelizumab (approximately 1 years).
  Other Names: SHR-1210

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Camrelizumab or Camrelizumab plus chemotherapy in patients with untreated, advanced ESCC with PD-L1 CPS≥10 ,who have been achieved PR and CR after treated with Camrelizumab.

DETAILED DESCRIPTION:
Standard 1L chemotherapy for advanced or metastatic esophageal squamous cell cancer(ESCC) results in poor OS(median<1year).Camrelizumab provided superior OS versus chemotherapy in heavily pretreated advanced/rucurrent ESCC.PD-1 antibody +chemo showed promisng antitumor activity in 1L advanced or metastatic ESCC.PD-L1 expression by CPS at cutoff≥10 has shown better enrichment for efficacy fo checkpoint inhibitors in ESCC.Recently, two clinical trials on Pembrolizumb have attracted our attention,KEYNOTE-181 and KEYNOTE-590.The median duration of response was 9.3 months in pembrolizumab monotherapy (KEYNOTE-181) ,and 8.3 months in Pembrolizumb plus chemotherapy (KEYNOTE-590). We hypothesis that administration of the PD-1 inhibitor will significantly prolong survival compared to PD-1 inhibitor combined with chemotherapy, when used as maintenance therapy in patients sensitive to PD-1 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female

  * Age ≥18 years
  * Histologically or cytologically confirmed locally advanced unresectable or metastatic ESCC
  * Measurable disease per RECIST v1.1 assessed by the local investigator
  * ECOG performance status 0 or 1
  * Provide newly obtained (preferred) or archival tissue sample
  * Negative urine or serum pregnancy test within 72 h before randomization (females)
  * Willing to use an adequate method of contraception throughout the study and for 120 days after the last dose of study medication and up to 180 days after the last dose of cisplatin
  * Adequate hematologic function, defined as ANC ≥ 1500/μl,platelet count ≥ 100,000/μl and hemoglobin ≥ 9.0 g/dl or ≥5.6 mmol/l
  * Adequate renal function, defined as creatinine ≤ 1.5 × ULN or measured or calculated creatinine clearance ≥ 60 mL/min for those with creatinine levels 1.5 × ULN
  * Adequate hepatic function, defined as total bilirubin ≤1.5 × ULN, or direct bilirubin ≤ ULN for those with total bilirubin levels 1.5 × ULN, and ALT/AST levels ≤ 2.5 × ULN
  * Adequate coagulation function, defined as INR ≤ 1.5 × ULN unless the patient is receiving anticoagulant therapy as long as PT or aPTT is within the therapeutic range
  * Written informed consent

Exclusion Criteria:

* • Locally advanced esophageal carcinoma that is resectable or potentially curable with radiation therapy per local investigator

  * Previous therapy for advanced disease
  * Major surgery, open biopsy or significant traumatic injury within 28 days before randomization or anticipated need for major surgery during the study treatment period
  * Known additional malignancy that is progressing or requires active treatment (except for BCC or SCC of the skin, in situ cervical cancer, in situ breast cancer that has undergone potentially curative treatment and in situ or intramucosal pharyngeal cancer)
  * Known active CNS metastases and/or carcinomatous meningitis; patients with previously treated and radiologically stable brain metastases may be eligible
  * Active autoimmune disease that has necessitated systemic treatment (other than replacement therapy) in the past 2 years
  * Diagnosis of immunodeficiency, receiving chronic systemic steroid therapy 10 mg daily prednisone equivalent or any other form of immunosuppressive therapy within 7 days before the first dose of study treatment or history of organ transplant including allogeneic stem cell transplant
  * Active infection necessitating systemic therapy
  * History or current evidence of any condition, therapy or laboratory abnormality that might confound the study results or interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
DOR | Up to 12 months
  DOR was defined as the time from the first documented a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) to progressive disease (PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of ≥1 new lesions was also considered PD) as assessed using RECIST v1.1.Median DOR as assessed by blinded independent central review per RECIST 1.1 is presented for participants who receive Camrelizumab with or without chemotherapy for advanced esophageal squamous cell cancer with a PD-L1 CPS ≥10.

SECONDARY OUTCOMES:
PFS | Up to 12 months
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of ≥1 new lesions was also considered PD. Median PFS as assessed by blinded independent central review per RECIST 1.1 is presented for participants who receive Camrelizumab with or without chemotherapy for advanced esophageal squamous cell cancer with a PD-L1 CPS ≥10.
OS | Up to 24 months
  OS was defined as the time from randomization to death due to any cause. Median OS in participants who receive Camrelizumab with or without chemotherapy for advanced esophageal squamous cell cancer with a PD-L1 CPS ≥10.
ORR | Up to 12 months
  ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. The percentage of participants with SCC of the esophagus who experienced a CR or PR is presented.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Doctor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China